CLINICAL TRIAL: NCT00940940
Title: Safety and Immunogenicity of Live Attenuated Herpes Zoster Vaccine in Patients Undergoing Living Donor Kidney Transplantations
Brief Title: Safety and Immunogenicity of Zostavax Vaccine in Patients Undergoing Living Donor Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: DKUA-001
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2015-05

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Live attenuated herpes zoster vaccine (Experimental)
  Interventions: Biological: Zostavax (Live attenuated herpes zoster vaccine)
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo vaccine

INTERVENTIONS:
Biological: Zostavax (Live attenuated herpes zoster vaccine) — 0.6 mL subcutaneous
  Other Names: Zostavax
  Arms: Live attenuated herpes zoster vaccine
Biological: Placebo vaccine — 0.65 mL subcutaneous
  Arms: Placebo

SUMMARY:
Varicella zoster virus is part of the herpesvirus group and causes chickenpox in exposed individuals. The majority of the population is seropositive for this virus. Reactivation of varicella zoster virus occurs in up to 30% of the general population over 60 years old.

Solid organ transplant recipients receive lifelong immunosuppression drugs and are at great risk of reactivation of all herpesviruses including the varicella zoster virus regardless of age. The vaccine has been shown to be effective in preventing shingles in the general population. The investigators' purpose is to determine how well the vaccine works in patients on renal replacement therapy and post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Listed or will likely be listed for live donor kidney transplant within one month

Exclusion Criteria:

1. Previous receipt of Zostavax

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2013-08-26 (Actual); Study Completion 2013-09-23 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada